CLINICAL TRIAL: NCT02430077
Title: Phase 2 Study of Obeticholic Acid for Lipodystrophy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abhimanyu Garg (Other)
Responsible Party: Sponsor-Investigator, Abhimanyu Garg, PROFESSOR, Internal Medicine, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU 062014-033
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Familial Partial Lipodystrophy
Keywords: Hepatic Steatosis
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Fatty Liver | interventions — obeticholic acid; Investigational New Drug Application

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active capsule of Obeticholic acid (Experimental): Patient will receive obeticholic acid (OCA) in the dose of 25 mg/day for a period of 4 months.
  Interventions: Drug: Obeticholic Acid
- Pacebo for Obeticholic acid (Placebo Comparator): Patient will recieve placebo in the dose of 25 mg/day for a period of 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid — Capsules of obeticholic acid (OCA) or an identical placebo in the dose of 25 mg/day for a period of 4 months .
  Other Names: NEW DRUG APPLICATION
  Arms: Active capsule of Obeticholic acid
Drug: Placebo — Identical to Obeticholic Acid - placebo drug
  Other Names: Identical to Obeticholic Acid placebo drug
  Arms: Pacebo for Obeticholic acid

SUMMARY:
Lipodystrophies are rare disorders characterized by selective loss of adipose tissue and predisposition to insulin resistance and its metabolic complications. Hepatic steatosis is a common complication in patients with partial and generalized lipodystrophies.Despite aggressive management of diabetes and hyperlipidemia, hepatic steatosis and its complications present a therapeutic challenge in many patients. Due to this large disease burden, it is important to assess the efficacy and safety of novel therapies for hepatic steatosis in patients with lipodystrophies.There are, however, no systematic studies evaluating various therapeutic interventions for reducing hepatic steatosis in patients with lipodystrophies. A variety of drugs have been investigated in nonlipodystrophic patients with non-alcoholic hepatic steatosis and steatohepatitis (NASH) or non-alcoholic fatty liver disease (NAFLD). Recent data support the activation of the farnesoid X receptor (FXR, NR1H4), a nuclear hormone receptor regulated by bile acids, for treatment of NASH and NAFLD. FXR activates transcription of several genes particularly the atypical nuclear receptor small heterodimer partner (SHP, NR0B2) and thus can influence triglyceride metabolism within hepatocytes.Both cholic acid (CA) and chenodeoxycholic acid (CDCA) are ligands for FXR, however, UDCA which is the 7 hydroxy β-epimer of CDCA, does not activate FXR. Obeticholic acid (OCA) is a first-in-class selective FXR agonist which has approximately 100 fold greater FXR-agonistic activity in the nanomolar range, as compared to CDCA .It therefore appears that FXR modulation offers interesting therapeutic possibilities in treating hepatic steatosis. This study is primarily designed to study efficacy of OCA, a strong FXR ligand, in reducing hepatic triglyceride levels in patients with hepatic steatosis and Familial Partial Lipodystrophy (FPLD). If proven to be effective, it may reduce morbidity and mortality as a result of sequelae of hepatic steatosis in patients with lipodystrophies.

DETAILED DESCRIPTION:
This study will be a randomized, placebo-controlled cross-over trial. Patients who are considered eligible for the study will undergo screening evaluation to determine their eligibility for the trial. For those who are found to be eligible, during the baseline period, they will continue their usual diet and other lifestyle measures without changing any medications for 1 month in order to establish a baseline state. Three blood samples will be obtained during this period at the Clinical and Translational Research Center. Following the baseline period, the patients will receive obeticholic acid (OCA) or an identical placebo in the dose of 25 mg/day for a period of 4 months and then will receive the other treatment (OCA or placebo) for 4 months. There will be a wash-out period of 4 months in-between the two study periods.

Patients will be educated to maintain their usual physical activities and diet during the study. The subjects will be admitted to the Clinical and Translational Research Center for the baseline evaluations (at the beginning of the two study periods), and at the end of four months during each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with familial partial lipodystrophy of the Dunnigan variety with heterozygous disease-causing missense mutation in lamin A/C (LMNA) gene.
2. Hepatic steatosis (>5.6% hepatic triglyceride content) as demonstrated by 1H magnetic resonance spectroscopy.
3. Age 18-70 years.
4. Alcohol intake of less than 20 g per day in females and 30 g per day in males.
5. Participants and their partners with whom they are having sex, must use medically-acceptable birth control (contraceptives) during the study. Medically-acceptable methods of contraception include: (1) surgical sterilization, such as hysterectomy, tubal ligation or vasectomy. (2) approved hormonal contraceptives, such as birth control pills, patch or ring; Depo-Provera, Implanon. (3) barrier methods, such as condom, cervical cap or diaphragm used with a spermicide. (4) an intrauterine device (IUD).

Exclusion Criteria:

1. Laboratory or other histologic findings highly suggestive of liver disease due to causes other than non-alcoholic steatohepatitis, such as chronic viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, biliary obstruction or genetic liver diseases such as Wilson's disease, hemochromatosis or alpha-1-antitrypsin deficiency.
2. Treatment with drugs associated with steatohepatitis, e.g., corticosteroids, high dose estrogens, methotrexate, amiodarone, tamoxifen, valproic acid, sulfasalazine, or oxacillin for more than 2 weeks in the 6 months prior to the study.
3. Decompensated liver disease as evidenced by clinical features of hepatic failure (variceal bleeding, ascites, hepatic encephalopathy etc.) and laboratory investigations (prolonged prothrombin time with INR > 1.3, hypoalbuminemia with serum albumin less than 3.0 g/dL, direct bilirubin > 1.3 mg/dL, or presence of esophageal varices etc.)
4. Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study suggestive of liver cancer.
5. Use of drugs which can potentially decrease hepatic steatosis during previous 3 months; ursodeoxycholic acid, thiazolidinediones, high-dose vitamin E, betaine, acetylcysteine and choline.
6. Significant systemic or major illnesses other than liver disease, such as congestive heart failure, cerebrovascular disease, respiratory failure, renal failure (serum creatinine >2 mg/dL), acute pancreatitis, organ transplantation, serious psychiatric disease, and malignancy, that could interfere with the trial and adequate follow up.
7. Acute medical illnesses precluding participation in the studies.
8. Known HIV-infected patient.
9. Current substance abuse.
10. Pregnant or lactating woman.
11. Hematocrit of less than 30%.
12. History of weight loss during past 3 months.
13. Patients on bile acid binding resins, cholestyramine, colestipol or colesevelam.
14. Hypersensitivity or intolerance to OCA or any components of its formulation.
15. Failure to give informed consent 16 .Previous clinical diagnosis of diabetes mellitus or fasting blood glucose ≥ 126 mg/dL or hemoglobin A1c ≥ 6.5%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT Southwestern Medical Center 5323 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of thirteen subjects were consented in the study. Ten adult female subjects completed the study. Two subjects did not qualify based on the enrollment criteria (screen failed). One subject withdrew due to personal reasons prior to being randomized. Hence only 10 subjects considered enrolled.
Groups:
- Active Capsule of Obeticholic Acid, Then Placebo: Patient received obeticholic acid (OCA) in the dose of 25 mg/day for a period of 4 months.
  Then a washout period of 4 months.
  Afterwards, patients received identical placebo in the dose of 25 mg/day for a period of 4 months .
- Placebo for Obeticholic Acid, Then Active Drug: Patient received placebo in the dose of 25 mg/day for a period of 4 months.
  Washout period of 4 months
  Thereafter, patients received Obeticholic Acid in the dose of 25 mg/day for a period of 4 months.
Period: First Intervention 4 Months
Arm/Group | Active Capsule of Obeticholic Acid, Then Placebo | Placebo for Obeticholic Acid, Then Active Drug
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout 4 Months
Arm/Group | Active Capsule of Obeticholic Acid, Then Placebo | Placebo for Obeticholic Acid, Then Active Drug
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention 4 Months
Arm/Group | Active Capsule of Obeticholic Acid, Then Placebo | Placebo for Obeticholic Acid, Then Active Drug
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of thirteen subjects were consented in the study. Ten adult female subjects completed the study. Two subjects did not qualify based on the enrollment criteria (screen failed). One subject withdrew due to personal reasons prior to being randomized. Hence only 10 subjects considered enrolled.
  Population Description: Baseline Characteristics of 10 patients
Groups:
- All Study Participants: Patients were randomized to receive Obeticholic acid or identical placebo in the dose of 25 mg/day for a period of 4 months. This was followed by a wash out period of 4 months. Thereafter, they crossed-over to receive Obeticholic acid or identical placebo in the dose of 25 mg/day for a period of 4 months.
  Placebo: Identical to Obeticholic Acid - placebo drug
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Liver Fat [Mean (Standard Deviation); unit: percentage of liver fat] | 13 (8)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Liver Triglycerides (TG).
Description: The primary end-point variable was the change in the liver TG content assessed using proton-density fat fraction mapping by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline, 4 months
Measure: Median (Full Range); unit: percentage of liver triglycerides
Groups:
- Baseline (Month 0): Before starting the active drug, Obeticholic Acid.
- Obeticholic Acid (Month 4): Patient recieved Obeticholic Acid in the dose of 25 mg/day for a period of 4 months.
- Placebo (Month 0): Before starting the Placebo
- Placebo (Month 4): Patient received placebo in the dose of 25 mg/day for a period of 4 months.
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of liver triglycerides | 13.2 [2.8 to 28.5] | 6.4 [2.4 to 18.0] | 12.3 [3.6 to 33.3] | 10.6 [3.4 to 29.3]

2. Secondary Outcome: Change in Serum Triglyceride Levels
Description: Change in the serum levels of Triglycerides from baseline to month 4 is being assessed.
Time Frame: Baseline, Month 4
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 10 | 10 | 10 | 10
mg/dL | 199.2 [78 to 392] | 182.3 [102 to 309.3] | 169.3 [103.5 to 562.0] | 161.3 [93 to 655]

3. Secondary Outcome: Change in Serum Levels of Alanine Aminotransferase
Description: Change in serum levels of Alanine Aminotransferase from baseline to month 4 is assessed
Time Frame: Baseline, Month 4
Measure: Median (Full Range); unit: U/L
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 10 | 10 | 10 | 10
U/L | 16.3 [13.5 to 31] | 15.8 [13 to 42.5] | 19.0 [11 to 33.5] | 18.5 [12.6 to 33]

4. Secondary Outcome: Change in Serum Levels of Aspartate Aminotransferases
Description: Change in serum levels of Aspartate Aminotransferases from baseline to month 4 is assessed
Time Frame: Baseline, Month4
Measure: Median (Full Range); unit: U/L
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 10 | 10 | 10 | 10
U/L | 15.5 [13.5 to 35.5] | 16.8 [13.7 to 27] | 18.7 [13.5 to 28.5] | 16.5 [12.5 to 31]

5. Secondary Outcome: Change in Serum Levels of Gamma-Glutamyl Transpeptidase
Description: Change in serum levels of Gamma-Glutamyl Transpeptidase from baseline to month 4 is assessed
Time Frame: Baseline, Month 4
Measure: Median (Full Range); unit: U/L
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 10 | 10 | 10 | 10
U/L | 27.5 [16.3 to 64] | 17 [10.6 to 45.7] | 21.6 [14.6 to 109] | 21.2 [13.5 to 66]

6. Secondary Outcome: Changes in Serum Insulin Levels
Description: Changes in serum Insulin levels is assessed
Time Frame: Baseline, Month 4
Population: Data was not collected
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Hepatic Insulin Sensitivity
Description: Change in hepatic insulin sensitivity is assessed by suppression of hepatic glucose output during the low-dose and high-dose insulin infusions during the euglycemic clamp study.
Time Frame: Baseline, Month 4
Population: Data not collected.
Arm/Group | Baseline (Month 0) | Obeticholic Acid (Month 4) | Placebo (Month 0) | Placebo (Month 4)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months for each intervention separated by a 4-month washout period, approximately 12 months total
Groups:
- Active Capsule of Obeticholic Acid: Patient received obeticholic acid (OCA) in the dose of 25 mg/day for a period of 4 months.
  Obeticholic Acid: Capsules of obeticholic acid (OCA) in the dose of 25 mg/day for a period of 4 months .
- Placebo for Obeticholic Acid: Patient received placebo in the dose of 25 mg/day for a period of 4 months.
  Placebo: Identical to Obeticholic Acid - no active ingredient
Arm/Group | Active Capsule of Obeticholic Acid | Placebo for Obeticholic Acid
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Capsule of Obeticholic Acid (N=10) | Placebo for Obeticholic Acid (N=10)
Itching (Skin and subcutaneous tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02430077/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02430077/ICF_001.pdf